CLINICAL TRIAL: NCT07048470
Title: Efficacy of Synbiotic Supplementation on IL-10, TGF-B and Disease Activity in Systemic Lupus Erythematosus Patients; A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy of Synbiotic Supplementation on IL-10, TGF-B and Disease Activity in Systemic Lupus Erythematosus Patients
Acronym: ESSENTIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Responsible Party: Principal Investigator, Yuniza, Principal investigator, Division of Allergy Immunology Faculty Member, Department of Internal Medicine, Universitas Sriwijaya/Mohammad Hoesin General Hospital, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DP.04.03/D.XVIII.6.8/ETIK/163
Record Dates: First submitted 2025-06-20; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; SLE; synbiotics; disease activity; MEX-SLEDAI; IL-10; TGF-β
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Synbiotics

STUDY DESIGN:
Intervention Model Description: This research is a double blind randomized controlled trial study. The study subjects were 36 patients diagnosed with mild to moderate lupus activity, randomly divided into 2 groups, who received synbiotic supplementation once daily for 12 weeks and the group that received placebo. Serum IL-10, TGF-β levels and the degree of disease activity using MEX-SLEDAI score were measured before and after treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Synbiotic (Experimental): The patients were given a capsule containing synbiotic once a day
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator): The patients were given placebo capsules once a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — The patients received synbiotics (containing Lactobacillus helveticus R0052 60%, Bifidobacterium infantis R0033 20%, Bifidobacterium bifidum R0071 20% and frukto-oligosaccharide 80 mg) supplementation
  Arms: Synbiotic
Dietary Supplement: Placebo — Patients received placebo capsules
  Arms: Placebo

SUMMARY:
Dysregulation of normal flora leads to dysbiosis, which has recently been investigated as an important internal environmental factor and has been proven to be associated with both active and remission phases of SLE, and can be used to predict disease activity. Administration of synbiotics is expected to restore mucosal barrier function and create an anti-inflammatory environment in the gut, by suppressing pro-inflammatory factors and increasing anti-inflammatory factors (IL-10 and TGF-β), leading to improved disease activity in SLE patients.

DETAILED DESCRIPTION:
This research is a double blind randomized controlled trial study. The study subjects were 36 patients diagnosed with mild to moderate lupus activity, randomly divided into 2 groups, who received synbiotic supplementation once daily for 12 weeks and the group that received placebo. Serum IL-10 and TGF-β levels and the degree of disease activity using MEX-SLEDAI score were measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria

1. All patients diagnosed with mild to moderate Systemic Lupus Erythematosus (SLE).
2. Patients aged over 18 years.
3. Willing to participate in the study by signing an informed consent form.
4. Have not consumed yogurt or supplements containing probiotics, prebiotics, or synbiotics within the last 2 weeks.

Exclusion Criteria

1. Severe SLE. 2, Pregnant or breastfeeding. 3. History of allergy to probiotics or prebiotics. 4. Patients with other immune-related disorders, whether autoimmune or immunocompromised conditions such as HIV or rheumatoid arthritis.

5. SLE with pulmonary tuberculosis. 6. Currently undergoing antibiotic therapy. 7. SLE with malignancy.

Drop-Out Criteria

1. Patients discontinue synbiotic intake for more than 2 weeks.
2. Death.
3. Occurrence of serious adverse drug reactions requiring discontinuation of the study drug.
4. Patients consume yogurt or supplements containing probiotics/synbiotics more than once per week outside of the study intervention, or undergo changes in steroid-sparing agents during the study period.
5. Patients require hospitalization due to symptom exacerbation during the intervention period.
6. Loss to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
IL-10 | From enrollment to the end of the treatment at 12 weeks
  To determine the effectiveness of adding synbiotics compared to placebo on IL-10 concentration change in Systemic Lupus Erythematosus Patients
TGF-B | From enrollment to the end of the treatment at 12 weeks
  To determine the effectiveness of adding synbiotics compared to placebo on TGF-B concentration change in Systemic Lupus Erythematosus Patients
MEX-SLEDAI score | From enrollment to the end of the treatment at 12 weeks
  To determine the effectiveness of adding synbiotics compared to placebo towards MEX-SLEDAI score changes

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Hoesin General Hospital, Palembang, South Sumatera, Indonesia

REFERENCES:
- [Background] Widhani A, Djauzi S, Suyatna FD, Dewi BE. Changes in Gut Microbiota and Systemic Inflammation after Synbiotic Supplementation in Patients with Systemic Lupus Erythematosus: A Randomized, Double-Blind, Placebo-Controlled Trial. Cells. 2022 Oct 29;11(21):3419. doi: 10.3390/cells11213419. PMID 36359816
- [Background] Askari G, Ghavami A, Shahdadian F, Moravejolahkami AR. Effect of synbiotics and probiotics supplementation on autoimmune diseases: A systematic review and meta-analysis of clinical trials. Clin Nutr. 2021 May;40(5):3221-3234. doi: 10.1016/j.clnu.2021.02.015. Epub 2021 Feb 17. PMID 33642142